CLINICAL TRIAL: NCT06332755
Title: A Phase 1a/1b, First-in-Human, Open-Label, Multi-Center, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LB-LR1109, When Administered Alone for the Treatment of Advanced or Metastatic Solid Tumors, and in Combination With Atezolizumab for the Treatment of Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study to Evaluate LB-LR1109, Administered Alone for the Treatment of Solid Tumor and in Combination With Atezolizumab for the Treatment of NSCLC
Acronym: LB-LR1109
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LG-LRCL001
Record Dates: First submitted 2024-02-16; First posted 2024-03-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer(NSCLC); Head and Neck Squamous Cell Carcinoma(HNSCC); Renal Cell Carcinoma(RCC); Urothelial Carcinoma; Malignant Melanoma
Keywords: solid tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Melanoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- phase 1a: Dose escalation / LB-LR1109 monotherapy (Experimental)
  Interventions: Drug: Phase 1a: LB-LR1109
- Phase 1b: Dose escalation / LB-LR1109 in combination with Atezolizumab (Experimental)
  Interventions: Drug: Phase 1b: LB-LR1109 and Atezolizumab

INTERVENTIONS:
Drug: Phase 1a: LB-LR1109 — intravenous administration
  Arms: phase 1a: Dose escalation / LB-LR1109 monotherapy
Drug: Phase 1b: LB-LR1109 and Atezolizumab — intravenous administration
  Arms: Phase 1b: Dose escalation / LB-LR1109 in combination with Atezolizumab

SUMMARY:
This is a Phase 1a/1b, first-in-human (FIH), multi-center, open-label, non-randomized, dose escalation study, designed to determine the Maximum tolerated dose(MTD)/Recommended Phase 2 dose (RP2D) and to evaluate safety, tolerability, preliminary efficacy, pharmacokinetics, immunogenicity, pharmacodynamics of LB-LR1109 as monotherapy in participants with advanced and/or metastatic non small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), renal cell carcinoma (RCC), urothelial carcinoma, or malignant melanoma and no available standard of care treatment options, and as combination therapy with atezolizumab in participants with advanced and/or metastatic NSCLC.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥18 years old at the time of signing the ICF.
2. (Phase 1a only) Participants must have 1 of the following histologically confirmed advanced or metastatic solid tumors with measurable or non-measurable disease as determined by RECIST v1.1,

   - NSCLC, HNSCC, RCC, urothelial carcinoma, or malignant melanoma.
3. (Phase 1a only) Participants who have metastatic disease which has progressed during or after approved standard therapies or are intolerant to approved therapies, or for which the participant refuses or is ineligible for standard therapy.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.
5. Life expectancy ≥12 weeks.
6. Participants with adequate organ function
7. No potential for childbearing or agree to use adequate contraception
8. Ability to understand the study purpose and procedures and have the willingness to sign a written informed consent document.
9. (Phase 1b only ) Must have histologically confirmed advanced or metastatic NSCLC without actionable genomic alteration that have approved therapies in the location where the participant's live and with measurable disease as determined by RECIST v1.1

Key Exclusion Criteria:

1. Clinically significant cardiac disease or cardiac failure.
2. Untreated or unstable brain or central nervous system (CNS) metastases or Leptomeningeal disease
3. Participants with any concurrent active malignancies
4. Has received prior therapy targeting LILRB or immunoglobulin-like transcript pathway.
5. History of life-threatening toxicity related to prior immune therapy
6. Has not recovered to ≤ Grade 1 or baseline from AEs and/or complications from prior surgical intervention or any anti-cancer treatment before starting study treatment
7. Participants must not have an active, known, or suspected autoimmune disease.
8. Evidence of active infection requiring IV antibiotic treatment ≤7 days prior to initiation of study treatment therapy (does not apply to viral infections that are presumed to be associated with the underlying tumor type required for study entry).
9. Pregnant or lactating or expecting to conceive a child during the study or within 6 months after the last dose of study intervention.
10. Any condition that would, in the Investigator's judgment, interfere with full participation in the study, including administration of study intervention and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
11. (Phase 1b only) Participants who were previously exposed to atezolizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: MTD and/or RP2D of LB-LR1109 as monotherapy in participants with advanced or metastatic solid tumors / Phase 1b: MTD and/or RP2D of LB-LR1109 as combination therapy with atezolizumab in participants with advanced or metastatic NSCLC | through study completion, an average of 1year
  Number of participants with dose-limiting toxicities (DLTs)
Phase 1a: Incidence of Treatment-Emergent Adverse Events of LB-LR1109 as monotherapy / Phase 1b: Incidence of Treatment-Emergent Adverse Events of LB-LR1109 as combination therapy with atezolizumab | through study completion, an average of 1year
  Incidence, severity (assessed by NCI CTCAE v5.0), and causality of AEs

SECONDARY OUTCOMES:
Phase 1a / 1b: Preliminary efficacy of LB-LR1109 as monotherapy and as combination therapy with atezolizumab | through study completion, an average of 1year
  ORR(overall response rate) assessed by RECIST v1.1 (%)
Phase 1a / 1b: Antitumor efficacy of LB-LR1109 as monotherapy and as combination therapy with atezolizumab | through study completion, an average of 1year
  PFS(Progression free survival)
Phase 1a/1b: Antitumor efficacy of LB-LR1109 as monotherapy and as combination therapy with atezolizumab | through study completion, an average of 1year
  OS (Overall survival) (months)
Phase 1a / 1b: Pharmacokinetic profile of LB-LR1109 as monotherapy and as combination therapy with atezolizumab | through study completion, an average of 1year
  Cmax (Maximum serum drug concentration)
Phase 1a / 1b: Characterize PK of LB-LR1109 as monotherapy and as combination therapy with atezolizumab | through study completion, an average of 1year
  Area under the concentration-time curve (AUC) 0-last
Phase 1a / 1b: Immunogenicity of LB-LR1109 as monotherapy and as combination therapy with atezolizumab | through study completion, an average of 1year
  Number and percentage of participants with ADAs

CONTACTS AND LOCATIONS:
Locations (1):
- NEXT Oncology, Fairfax, Virginia, United States